CLINICAL TRIAL: NCT05197153
Title: A Phase II, Prospective, Randomized, Observer-blinded, Multi-Center Study to Evaluate the Safety, Tolerability, and Immunogenicity of Heterologous Booster Dose With AZD1222, mRNA-1273, or MVC-COV1901 COVID-19 Vaccine in Adults
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Booster With AZD1222, mRNA-1273, or MVC-COV1901 Against COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CT-COV-24
Record Dates: First submitted 2021-12-13; First posted 2022-01-19 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Vaccine
Keywords: COVID-19 Vaccine
MeSH Terms: interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Half dose of MVC-COV1901 (Experimental): 7.5 mcg of S-2P protein with adjuvant
  Interventions: Biological: Half dose of MVC-COV1901
- Full dose of MVC-COV1901 (Experimental): 15 mcg of S-2P protein with adjuvant
  Interventions: Biological: Full dose of MVC-COV1901
- AZD1222 (Experimental): 5*10^10 viral particles of AZD1222
  Interventions: Biological: AZD1222
- Half dose of mRNA-1273 (Active Comparator): 50 mcg mRNA encoding the pre-fusion stabilized S protein
  Interventions: Biological: Half dose of mRNA-1273

INTERVENTIONS:
Biological: Half dose of MVC-COV1901 — Approximately 240 participants will receive 1 doses of half of MVC-COV1901(S-2P protein with adjuvant) at Visit 2 (Day 1) via intramuscular (IM) injection in the deltoid region.
  Arms: Half dose of MVC-COV1901
Biological: Full dose of MVC-COV1901 — Approximately 240 participants will receive 1 doses of MVC-COV1901(S-2P protein with adjuvant) at Visit 2 (Day 1) via intramuscular (IM) injection in the deltoid region.
  Arms: Full dose of MVC-COV1901
Biological: AZD1222 — Approximately 240 participants will receive 1 doses of AZD1222 at Visit 2 (Day 1) via intramuscular (IM) injection in the deltoid region.
  Arms: AZD1222
Biological: Half dose of mRNA-1273 — Approximately 240 participants will receive 1 doses half of mRNA-1273 at Visit 2 (Day 1) via intramuscular (IM) injection in the deltoid region.
  Arms: Half dose of mRNA-1273

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of booster dose of vaccine in participants who are generally healthy or with stable pre-existing health conditions. Study details include:

* The study duration per participant will be approximately 209 days (28 days screening, 1 day vaccination, and 180 days follow-up).
* The treatment will include 1 booster dose only.
* The visit frequency will be 6 on-site visits and 1 phone visit.

DETAILED DESCRIPTION:
This is a Phase II, prospective, randomized, observer-blinded, multi-center study, to evaluate the safety, tolerability, and immunogenicity of a booster vaccination with AZD1222, mRNA-1273, or MVC-COV1901 vaccine. Approximately 960 participants aged 18 ~ < 80 years, who received homologous two doses of vaccines 150 ~ 365 days ago, will be enrolled and divided into three groups. Each group will consist of 320 eligible subjects, and for each group the randomization will be stratified according to study site and age to four treatments (AZD1222, half dose of mRNA-1273, full dose or half dose of MVC-COV1901 in 1:1:1:1 ratio). Therefore, within a group, for either age stratum, there will be at least 30 participants for each treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥ 18 years at randomization.
2. Healthy adults or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease 3 months before enrollment and expected to remain stable for the duration of the study.
3. Documented to have received two homologous doses of AZD1222, mRNA-1273, or MVC-COV1901 vaccine, with the latest dose between 150 and 365 days prior to randomization, with an interval between the two homologous doses of ≥ 4 weeks to ≤ 12 weeks, and did not receive any other investigational or approved COVID-19 vaccines
4. Female participants must:

   1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following the injection of study intervention. Acceptable forms include:

   i.Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii.Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository c.Have a negative pregnancy test
5. Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
6. Participant, and the participant's legal representative if applicable, must understand the procedures of the study and provide written informed consent.

Exclusion Criteria:

1. Pregnant or breast feeding or have plan to become pregnant in 30 days after the administration of study intervention.
2. Employees at the investigator's site, of the Sponsor or delegate (e.g., contract research organization) who are directly involved in the conduct of the study.
3. Currently receiving or received any investigational intervention within 30 days prior to the vaccination of study intervention.
4. Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live-attenuated vaccines within 7 days prior to vaccination of study intervention.
5. Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the vaccination of study intervention.
6. Currently receiving or anticipated to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the vaccination of study intervention.
7. Currently receiving or anticipated to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks prior to the vaccination of study intervention.
8. Major surgery or any radiation therapy within 12 weeks prior to the vaccination of study intervention.
9. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
10. A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
11. Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
12. A history of cerebral venous sinus thrombosis, heparin-induced thrombocytopenia, thrombosis with thrombocytopenia syndrome (TTS), antiphospholipid syndrome, capillary leak syndrome, myocarditis, or pericarditis
13. Participant with ongoing acute diseases or serious medical conditions which will interfere with adherence to study requirements, or the evaluation of any study endpoint.

    Acute diseases or serious medical conditions include cardiovascular, pulmonary, hepatic, neurologic, metabolic, renal, psychiatric condition (e.g. alcoholism, drug abuse, anorexia or severe depression), current severe infections, autoimmune disease, medical history, physical findings, or laboratory abnormality that in the investigators' opinion are not in stable condition and participating in the study could adversely affect the safety of the participant.
14. Documented SARS-CoV1 or 2 infection prior to the study intervention.
15. Participant with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the AZD1222, mRNA-1273 or MVC-COV1901.
16. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the vaccination of study intervention.
17. Any condition that is a contraindication to study intervention based on the judgement of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events from Day 1 to 28 | Day1 to 28 days after vaccination
  To measure the incidence of adverse event from Day 1 to Day 28 after the booster dose.
  * Solicited local adverse events (AEs) (up to 7 days after injection of booster dose)
  * Solicited systemic AEs (up to 7 days after injection of booster dose)
  * Unsolicited AEs (up to 28 days after injection of booster dose)
  * AE of special interest (AESI)
  * Vaccine-associated enhanced disease (VAED)
  * Serious adverse event (SAE)
Primary Immunogenicity-1 | Day1 to Day 29
  To evaluate the immunogenicity in terms of Anti-SARS-CoV-2 neutralizing antibody at Day 29
  • GMT
Primary Immunogenicity-2 | Day1 to Day 29
  To evaluate the immunogenicity in terms of Anti-SARS-CoV-2 neutralizing antibody at Day 29
  • Seroconversion rate (SCR)
Primary Immunogenicity-3 | Day1 to Day 29
  To evaluate the immunogenicity in terms of Anti-SARS-CoV-2 neutralizing antibody at Day 29
  • GMT ratio
Primary Immunogenicity-4 | Day1 to Day 29
  To evaluate the immunogenicity in terms of Anti-SARS-CoV-2 neutralizing antibody at Day 29
  • Seroresponse rate

SECONDARY OUTCOMES:
Incidence of Adverse Events from Day 1 to 181 | Day 1 to Day 181
  To measure the incidence of adverse event throughout the whole study period.
  * ≥ Grade 3 AE
  * AESI
  * VAED
  * SAE
Secondary Immunogenicity (Humoral)-1 | Day 1 to Day 181
  To evaluate the immunogenicity in terms of Anti-spike IgG
  • GMT
Secondary Immunogenicity (Humoral)-2 | Day 1 to Day 181
  To evaluate the immunogenicity in terms of Anti-spike IgG
  • SCR
Secondary Immunogenicity (Humoral)-3 | Day 1 to Day 181
  To evaluate the immunogenicity in terms of Anti-spike IgG
  • GMT ratio
Secondary Immunogenicity (Cellular) | Day 1 to Day 15
  To evaluate the cellular immunology by Enzyme-linked immunoSpot assay (ELISpot)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Lien, MD. DrPH, Study Chair — Medigen Vaccine Biologics
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - Taipei Veteran General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estephan L, Lin YC, Lin YT, Chen YH, Pan SC, Hsieh SM, Torkehagen PF, Weng YJ, Cheng HY, Estrada JA, Waits A, Chen C, Lien CE. Safety and immunogenicity of homologous versus heterologous booster dose with AZD1222, mRNA-1273, or MVC-COV1901 SARS-CoV-2 vaccines in adults: An observer-blinded, multi-center, phase 2 randomized trial. Vaccine. 2023 May 26;41(23):3497-3505. doi: 10.1016/j.vaccine.2023.04.029. Epub 2023 Apr 12. PMID 37080829